CLINICAL TRIAL: NCT02876185
Title: Evaluation of the Possibility to Delegate Glaucoma Surveillance to Orthoptists in Hospital
Acronym: GLAUS
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ICU_2015_39
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Glaucoma
Keywords: Glaucoma surveillance; Orthoptist
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with glaucoma: Patients presenting an open-angle glaucoma or ocular hypertension
  Interventions: Other: Monitoring by an orthoptist then by an ophthalmologist

INTERVENTIONS:
Other: Monitoring by an orthoptist then by an ophthalmologist — At each visit, the usual monitoring tests will be collected and viewed by the orthoptist then by the ophthalmologist concerning the necessity of an anticipated ophthalmological consultation

SUMMARY:
Glaucoma is a progressive optical neuropathy, generally associated with ocular hypertension. The treatment aims to stabilize the visual field deficiencies by lowering the intraocular pressure. Due to the fluctuation of the visual field test and re-test measures, the European recommendations are to obtain 6 visual field tests in 2 years (or one every 4 months) in order to know if the pathology is progressing despite the current treatment (or if the treatment is necessary, in cases of intraocular hypertensions). The lack of ophthalmologists renders the monitoring of a beginning glaucoma, rarely compatible with the present recommendations. It is therefore crucial to evaluate new therapeutic alternatives, when faced to a decreasing medical demography and an increase the patient's needs.

This study should allow to validate the possibility to delegate monitoring tasks to orthoptists during glaucoma surveillance. To organize the delegation of this surveillance to orthoptists would permit a better distribution of the ophthalmologist's activities.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years old or more
* Open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* Other active ocular pathology
* Monophthalmic patients
* Patients requiring a Goldmann visual field exam
* Opposition of the patient to participate to the trial
* Pregnant women or breastfeeding
* Patient under juridical protection
* Lack of affiliation to social security or universal health coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an open-angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
detection by the orthoptists of an abnormality that would require an anticipated ophthalmologic consultation | 20 month of follow-up

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre hospitalier, Angers
  - Hôpital Ambroise-Paré, Boulogne-Billancourt
  - Clinique Universitaire d'Ophtalmologie, Grenoble
  - Fondation Ophtalmologique A de Rothschild, Paris